CLINICAL TRIAL: NCT05962346
Title: Pilot Trial of Fetoscopic Endoluminal Tracheal Occlusion for Severe Left Congenital Diaphragmatic Hernia
Brief Title: Fetal Endoscopic Tracheal Occlusion for Congenital Diaphragmatic Hernia
Acronym: FETO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mauro H. Schenone (Other)
Responsible Party: Sponsor-Investigator, Mauro H. Schenone, Regulatory Sponsor and Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-002166
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2025-06-30 (Actual); Status verified 2025-04

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital | interventions — Fetoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- FETO Group (Experimental): Participants will undergo fetal endoscopic tracheal occlusion (FETO) surgical procedure between 27 weeks 0 days and 29 weeks 6 days gestation.
  Interventions: Device: BALT GOLDBALL 2 detachable latex ballon; Device: BALTACCIBDPE100 Microcatheter; Device: Storz fetoscopic operating sheath and miniature telescope/fetoscope

INTERVENTIONS:
Device: BALT GOLDBALL 2 detachable latex ballon — Inflated with fluid in the fetal trachea and provide with the occlusion necessary to promote lung growth.
Device: BALTACCIBDPE100 Microcatheter — Used to deliver the detachable balloon
Device: Storz fetoscopic operating sheath and miniature telescope/fetoscope — Used to percutaneously enter though the maternal abdominal wall, uterus and into the amniotic cavity, fetal mouth, pharynx, larynx, into the trachea where the delivery catheter will be used to deliver the detachable balloon that will provide with the tracheal occlusion.

SUMMARY:
The purpose of this research is to gather information on the safety and effectiveness of a procedure called Fetoscopic Endoluminal Tracheal Occlusion (FETO) at Mayo Clinic. The intent of the FETO procedure is to improve development of the lungs in fetuses diagnosed with severe congenital diaphragmatic hernia (CDH).

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Normal fetal karyotype or microarray. Results by fluorescence in situ hybridization (FISH) will be acceptable if the patient is > 26 weeks
* Isolated severe left CDH with O/E LHR < 25% )
* Gestation age at enrollment prior to 29 wks plus 6 days.
* Pulmonary hypoplasia with ultrasound O/E LHR < 25% (measured at 18 0/7 to 29 5/7 weeks) at the time of surgery.
* Gestational age at FETO procedure 27 weeks 0 days to 29 weeks 6 days as determined by clinical information (LMP) and evaluation of first ultrasound
* Patient meets psychosocial criteria: able to reside within 30 minutes of Mayo Clinic, Rochester and able to comply with the travel for the follow-up requirements of the trial; patient has a support person (e.g. spouse, partner, mother) available to stay with the patient for the duration of the pregnancy at Mayo Clinic
* Patient is willing and able to give informed consent
* Appropriate multi-disciplinary counseling performed with maternal-fetal medicine, neonatology, pediatric surgery, genetics, pediatric otolaryngology (ENT)

Exclusion Criteria:

* Multi-fetal pregnancy
* History of natural rubber latex allergy
* Preterm labor, cervix shortened (<20 mm) at enrollment or within 24 hours of FETO balloon insertion procedure) or uterine anomaly strongly predisposing to preterm labor
* Psychosocial ineligibility, precluding consent: inability to reside within 30 minutes of Mayo Clinic, Rochester and inability to comply with the travel for the follow-up requirements of the trial; patient does not have a support person (e.g. spouse, partner, mother) available to stay with the patient for the duration of the pregnancy at Mayo Clinic
* Right sided CDH or bilateral CDH, isolated left sided with O/E LHR >25% measured at 18 0/7 to 29 6/7 weeks) as determined by ultrasound
* Additional fetal anomaly and chromosomal abnormalities by ultrasound, MRI, or echocardiogram that will significantly worsen prognosis. No cases will be removed post hoc if abnormalities are discovered in the course of post-operative monitoring
* Maternal contraindication to fetoscopic surgery
* History of incompetent cervix with or without cerclage
* Placental abnormalities (previa, abruption, accreta) known at time of enrollment
* Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
* Maternal HIV, Hepatitis-B, Hepatitis-C status positive.
* Uterine anomaly such as large or multiple fibroids or mullerian duct abnormality that will make the procedure technically unfeasible
* No safe or technically feasible fetoscopic approach to balloon placement
* Participation in another intervention study that influences maternal and fetal morbidity and mortality or participation in this trial in a previous pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2043-07 (Estimated); Study Completion 2043-07 (Estimated)

PRIMARY OUTCOMES:
Technical success of the balloon placement procedure | Up to 29 weeks gestation
  The number of successful balloon placement procedures defined as balloon was correctly inflated and placed/secured in the trachea.
Technical success of balloon retrieval procedure | Up to 34 weeks gestation
  The number of successful balloon retrieval procedure defined as antenatal removal of the balloon.
Operative times | Up to 34 weeks gestation
  FETO placement and release operative times reported in minutes
Frequency of unplanned balloon removal | Up to 34 weeks gestation
  The frequency of non-emergent and emergent completion of FETO release (unplanned balloon removal)
Number of incidences of maternal complications | Up to 41 weeks gestation
  Maternal complications including preterm labor, premature rupture of membranes, oligohydramnios, polyhydramnios, chorioamnionitis
Gestational Age at Delivery | Up to 41 weeks gestation
  Gestation Age reported at time of delivery

SECONDARY OUTCOMES:
Fetal Lung Growth as measured via Fetal Lung Volume | Up to 24 months post partum
  Fetal Lung Volume as measured via ultrasound
Fetal Lung Growth as measured via LHR | Up to 24 months post partum
  Lung area to head circumference Ratio (LHR) as measured via ultrasound
Fetal Survival | Up to 6 months post partum
  Survival at 30 days, discharge from the hospital and at 6 months if still hospitalized
Fetal Oxygen Dependency | Up to 24 months post partum
  Oxygen dependency graded as none, mild, moderate, severe as assessed by treating physician
Occurrence of severe pulmonary hypertension | Up to 24 months post partum
  Number of occurrence of severe pulmonary hypertension in infants based on echocardiogram
ECMO Support | Up to 24 months post partum
  Number of infants reported that required Extracorporeal membrane oxygenation (ECMO) support
Number of days in NICU | Up to 24 months post partum
  Number of days infant was in neonatal intensive care unit
Number of days of ventilator support | Up to 24 months post partum
  Number of reported days infants required ventilator support
Number of periventricular leukomalacia at < 2 months postnatally | Up to 2 months post partum
  Number of infants reported presence of periventricular leukomalacia at < 2 months postnatally
Number of infant complications | Up to 24 months post partum
  Number of infants reporting the presence of: neonatal sepsis, intraventricular hemorrhage (grade 3 or higher), retinopathy of prematurity (grade 3 or higher) or gastro-esophageal reflux
Use of patch or muscle flap | Up to 24 months post partum
  Number of infants reported to require the use of patch or muscle flap
Maternal hospitalization | Up to 24 months post partum
  Number of reported days of maternal hospitalization
Route of delivery | Day 1 (post partum)
  Number of participants that delivered vaginally and via caesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Schenone, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials